CLINICAL TRIAL: NCT05011149
Title: Selective Early Medical Treatment of the Patent Ductus Arteriosus in Extremely Low Gestational Age Infants: A Pilot Randomized Controlled Trial
Brief Title: Selective Early Medical Treatment of Patent Ductus Arteriosus in Extremely Low Gestational Age Infants: A Pilot RCT
Acronym: SMART-PDA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: IWK Health Centre (Other)
Collaborators: BC Children's Hospital Research Institute (Other); CHU de Quebec-Universite Laval (Other); Sunnybrook Health Sciences Centre (Other); Mount Sinai Hospital, Canada (Other); Sharp Mary Birch Hospital for Women & Newborns (Other); Canadian Institutes of Health Research (CIHR) (Other Government); Dalhousie Medical Research Foundation (Unknown); Children's Hospital of Orange County, OC, California, United States (Unknown); University of Alberta (Other); University of Oklahoma (Other)
Responsible Party: Principal Investigator, Dr. Souvik Mitra, MD MSc FRCPC, Associate Professor & Neonatologist, IWK Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 459750
Record Dates: First submitted 2021-08-12; First posted 2021-08-18 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Patent Ductus Arteriosus After Premature Birth
Keywords: extremely preterm infant; early medical treatment; randomized controlled trial
MeSH Terms: interventions — Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Selective early medical treatment (SMART) strategy (Experimental): Infants who are randomized to experimental group will follow the SMART treatment protocol, which includes echocardiographic screening every 72 hours to categorize PDA disease severity by combining clinical and echocardiographic features. At any evaluation if patients are found to have a "severe PDA" on echocardiography, irrespective of clinical symptoms, or a "moderate PDA" on echocardiography with at least moderate clinical illness, they will receive pharmacotherapy aimed at PDA closure (The PDA severity has been divided into mild, moderate or severe based on pre-defined clinical and echocardiographic criteria).
  Interventions: Drug: Ibuprofen
- Early conservative management strategy (No Intervention): Infants randomized to this arm will not undergo any further echocardiographic assessment or pharmacological treatment of the PDA regardless of the clinical signs. If the infant gets an echocardiographic assessment for a reason different than PDA assessment (such as hypotension or oxygenation failure) and a PDA is incidentally noted that fits the treatment criteria, the infant will not be initiated on pharmacotherapy. After 7 days of age, decision on PDA assessment and treatment will be at the discretion of the treating physician.

INTERVENTIONS:
Drug: Ibuprofen — Pharmacotherapy, when indicated (ie, for "severe PDA" on echocardiography, irrespective of clinical symptoms, or a "moderate PDA" on echocardiography with at least moderate clinical illness), will be provided in the form of ibuprofen as first line agent at a standard dosing of 10 mg/kg followed by 2 doses of 5mg/kg every 24 h. The route of administration may be intravenous or enteral, as determined by the treating team.
  For treated infants, follow-up echocardiography will be conducted at the end of the 3-day course and second course of treatment will be initiated if they still fulfill study treatment criteria as mentioned above. If any treatment-eligible infant has a contraindication to ibuprofen, use of acetaminophen will be permitted as an alternative agent.
  Arms: Selective early medical treatment (SMART) strategy

SUMMARY:
Background: Among preterm infants, those born at a gestational age less than 26 weeks are considered the most vulnerable with a high risk of short- and long-term health problems that include chronic lung disease, brain bleeds, gut injury, kidney failure and death. Patent ductus arteriosus (PDA) is the most common heart condition with almost 70% preterm infants in this gestational age group being diagnosed with a PDA. Though many PDAs spontaneously resolve on their own, research suggests that if the PDA persists, it may contribute to a number of these short- and long-term health problems. Non-steroidal anti-inflammatory medications such as ibuprofen are commonly used to treat a PDA. Such drugs can also have harmful effects on the gut and kidneys of extremely preterm infants. Therefore, we are unsure if early treatment of a symptomatic PDA in this age group is at all beneficial. Given the wide variation in PDA treatment approaches in this age group, a randomized trial design, where extremely preterm infants with a symptomatic PDA are randomly assigned to early treatment or no early treatment, is essential to address this question.

Purpose of the study: The overall purpose of this pilot study is to assess the feasibility of conducting a large study to explore the following research question: In preterm infants born <26 weeks' gestation, is a strategy of selective early medical treatment of a symptomatic PDA better than no treatment at all in the first week of life?

The main feasibility objectives of this study are:

1. To assess how many eligible infants can be enrolled in the study
2. To assess how many enrolled infants properly complete the study protocol

Importance: To our knowledge this will be the first study on PDA management in preterm infants that specifically aims to enroll preterm infants born at <26 weeks of gestational age who are at the highest risk for PDA-related problems but have been mostly under-represented in previous PDA studies.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants less than 26 completed weeks (i.e., up to and including 25 weeks and 6 days) of gestation

Exclusion Criteria:

* no PDA on initial screening echocardiography
* congenital heart disease (excluding patent foramen ovale, atrial septal defect or ventricular septal defect with a defect size less than 2mm)
* other major congenital anomaly
* decision to withhold/withdraw care

Max Age: 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of eligible infants recruited during the study period | 7 days postnatal age
Proportion of randomized infants with no reported protocol deviations | 7 days postnatal age

SECONDARY OUTCOMES:
Proportion of infants in control group meeting pre-defined safety criteria | 7 days postnatal age
Reasons for non-recruitment | 7 days postnatal age
  qualitative description of reasons for non-recruitment of eligible infants
Reasons for non-adherence to protocol | 7 days postnatal age
  qualitative description of reasons for non-adherence to protocol in randomized infants
Completeness of data collection for clinical outcomes | through hospital discharge (approximately 20 weeks postnatal age unless death occurs first)
  Proportion of recruited infants with complete clinical outcome data
All-cause mortality during hospital stay | through hospital discharge (approximately 20 weeks postnatal age unless death occurs first)
Surgical/interventional PDA closure | through hospital discharge (approximately 20 weeks postnatal age unless death occurs first)
Receipt of any PDA pharmacotherapy | through hospital discharge (approximately 20 weeks postnatal age unless death occurs first)
Receipt of open-label rescue medical treatment in the control group | 7 days postnatal age
Chronic lung disease | birth through 36 weeks post menstrual age
  Oxygen or respiratory support requirement at 36 weeks' postmenstrual age or at discharge
Postnatal corticosteroid use | through hospital discharge (approximately 20 weeks postnatal age unless death occurs first)
Pulmonary hemorrhage | 7 days postnatal age
  blood-stained respiratory secretions with a significant increase in respiratory requirements (MAP>12 and/or FiO2>60%)
Duration of invasive mechanical ventilation | through hospital discharge (approximately 20 weeks postnatal age unless death occurs first)
  Number of days on mechanical ventilation with an endotracheal tube
Intraventricular hemorrhage | through hospital discharge (approximately 20 weeks postnatal age unless death occurs first)
  Grade I-IV according to Papile Criteria
Severe intraventricular hemorrhage | through hospital discharge (approximately 20 weeks postnatal age unless death occurs first)
  Grade III-IV according to Papile Criteria
Periventricular leukomalacia | through hospital discharge (approximately 20 weeks postnatal age unless death occurs first)
Necrotizing enterocolitis | through hospital discharge (approximately 20 weeks postnatal age unless death occurs first)
  Stage 2 or greater as per Bell's criteria
Gastrointestinal bleeding | within seven days of the first dose of pharmacotherapy
Gastrointestinal perforation | through hospital discharge (approximately 20 weeks postnatal age unless death occurs first)
Severe retinopathy of prematurity | through hospital discharge (approximately 20 weeks postnatal age unless death occurs first)
  stage 3 or greater
Definite sepsis | through hospital discharge (approximately 20 weeks postnatal age unless death occurs first)
  Clinical symptoms and signs of sepsis and a positive bacterial culture in a specimen obtained from normally sterile fluids or tissue obtained at postmortem
Oliguria | 7 days postnatal age
  urine output less than 1 mL/kg/hour
Duration of hospitalization (days) | through hospital discharge (approximately 20 weeks postnatal age unless death occurs first)

CONTACTS AND LOCATIONS:
Overall Officials: Souvik Mitra, MD, MSc, Principal Investigator — Dalhousie University & IWK Health
Locations (9):
- United States (3):
  - Children's Hospital of Orange County, Orange, California
  - Sharp Mary Birch Hospital for Women & Newborns, San Diego, California
  - OU College of Medicine, University of Oklahoma, Oklahoma City, Oklahoma
- Canada (6):
  - Stollery Children's Hospital, Edmonton, Alberta
  - British Columbia Women's Hospital, Vancouver, British Columbia
  - IWK Health Center, Halifax, Nova Scotia
  - Mount Sinai Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data on clinical outcomes collected during the trial will be shared after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: As soon as possible, wherever legally and ethically possible. In addition, data from the trial will be made available upon reasonable request.

REFERENCES:
- [Derived] Mitra S, Hebert A, Castaldo M, Disher T, El-Naggar W, Dhillon S, Alhassen Z, Koo J, Katheria AC, Hyderi A, Kumaran K, Makoni M, Weisz DE, Jain A, Bacchini F, Cameron A, Hatfield T, Dorling J, McNamara PJ, Thabane L. Selective early medical treatment of the patent ductus arteriosus in extremely low gestational age infants: a pilot randomised controlled trial protocol (SMART-PDA). BMJ Open. 2024 Jul 24;14(7):e087998. doi: 10.1136/bmjopen-2024-087998. PMID 39053961
- See also: Project funding information on the Canadian Institutes of Health Research (CIHR) Funding Decision Database — https://webapps.cihr-irsc.gc.ca/decisions/p/project_details.html?applId=441822&lang=en